CLINICAL TRIAL: NCT00419900
Title: Use of Hair to Diagnose the Presence of Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fermiscan Ltd (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: FER2k
Record Dates: First submitted 2007-01-07; First posted 2007-01-09 (Estimated); Last update posted 2007-01-09 (Estimated); Status verified 2007-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; diagnosis; x-ray diffraction; synchrotron; hair
MeSH Terms: conditions — Breast Neoplasms; Disease

INTERVENTIONS:
Procedure: diagnosis of breast cancer by x-ray diffraction of hair

SUMMARY:
Using synchrotron X-ray diffraction, it has been reported that a hair from an individual with breast cancer exhibits a difference in its molecular structure compared to that of an individual without breast cancer. This difference is visible in the X-ray diffraction pattern as a ring superimposed on the pattern for normal hair.

The hypothesis of this study is that synchrotron x-ray diffraction can be used to differentiate hairs from women with medically diagnosed breast cancer from women not known to have the disease.

To test this hypothesis, hair from 2000 women attending radiology clinics for mammography will be collected, analysed by x-ray diffraction and then analysed using Fermiscan proprietary image analysis software. The mammogram status of the subjects will be blinded from the diffraction analysts. Results will then be compared with mammography results to allow a direct comparison between the Fermiscan test and mammography in terms of specificity and sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (aged >20) who are undergoing mammography, and
* Who are willing and able to provide informed consent; and
* Who have usable scalp and/or pubic hair

Exclusion Criteria:

* Women who have dyed or permed their scalp hair within the previous 6 weeks and whose pubic hair is unavailable;
* Women with a history of breast cancer ever or other cancers (excluding non-melanoma skin cancer and CIN [cervical intra-epithelial neoplasia]) within 5 years.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000
Dates: Start 2006-12

PRIMARY OUTCOMES:
Accuracy (sensitivity and specificity) of the breast cancer test based on detection of an abnormal pattern of hair x-ray diffraction compared to the gold standard of mammography plus biopsy where indicated

SECONDARY OUTCOMES:
The prevalence of a positive hair x-ray diffraction pattern and a negative mammogram; and the prevalence of a negative hair x-ray diffraction pattern and a positive mammogram;

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Yuile, MBBS, FRACR, Principal Investigator — Radiation Oncology Associates, Sydney, Australia
Locations (5):
- Australia (5):
  - Bankstown Diagnostic Imaging Centre, Sydney, New South Wales
  - Campbelltown Ultrascan Radiology, Sydney, New South Wales
  - Diagnostic Imaging Centre, St George Private Hospital, Sydney, New South Wales
  - Liverpool Ultrascan Radiology, Sydney, New South Wales
  - Penrith Imaging, Sydney, New South Wales

REFERENCES:
- [Background] James VJ. A place for fiber diffraction in the detection of breast cancer? Cancer Detect Prev. 2006;30(3):233-8. doi: 10.1016/j.cdp.2006.04.001. Epub 2006 Jul 28. PMID 16876335
- [Background] James V, Corino G, Robertson T, Dutton N, Halas D, Boyd A, Bentel J, Papadimitriou J. Early diagnosis of breast cancer by hair diffraction. Int J Cancer. 2005 May 10;114(6):969-72. doi: 10.1002/ijc.20824. PMID 15645416
- [Background] James V. False-positive results in studies of changes in fiber diffraction of hair from patients with breast cancer may not be false. J Natl Cancer Inst. 2003 Jan 15;95(2):170-1. doi: 10.1093/jnci/95.2.170. No abstract available. PMID 12529353
- [Background] Meyer P, James VJ. Experimental confirmation of a distinctive diffraction pattern in hair from women with breast cancer. J Natl Cancer Inst. 2001 Jun 6;93(11):873-5. doi: 10.1093/jnci/93.11.873. No abstract available. PMID 11390537
- [Background] James V, Kearsley J, Irving T, Amemiya Y, Cookson D. Using hair to screen for breast cancer. Nature. 1999 Mar 4;398(6722):33-4. doi: 10.1038/17949. No abstract available. PMID 10078527